CLINICAL TRIAL: NCT06538519
Title: Gait Analysis and Clinical Outcomes of Anterior and Lateral Approach Total Hip Arthroplasty. A Prospective Randomized Study.
Brief Title: Gait Analysis and Clinical Outcomes of Anterior and Lateral Approach Total Hip Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MD 03/2021
Record Dates: First submitted 2024-07-07; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Hip Osteoarthritis
Keywords: arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct anterior approach group (Active Comparator)
  Interventions: Procedure: total hip replacement using anterior approach; Device: gait analysis at 6wks, 3 months and 18 months
- lateral approach group (Active Comparator)
  Interventions: Procedure: total hip replacement using lateral approach; Device: gait analysis at 6wks, 3 months and 18 months

INTERVENTIONS:
Procedure: total hip replacement using lateral approach — In the lateral approach partial detachment of the anterior one-third of the gluteus medius muscle.
  Arms: lateral approach group
Procedure: total hip replacement using anterior approach — the anterior approach using an internervous plane between the tensor fascia latae and the sartorius muscle.
  Arms: direct anterior approach group
Device: gait analysis at 6wks, 3 months and 18 months — gait analysis done in the gait lab at the mentioned postoperative periods

SUMMARY:
The goal of this Prospective Randomized Study is to confirm presence or absence of differences in gait mechanics in direct anterior and lateral approaches for total hip arthroplasty. and to compare the clinical outcomes of both approaches.

The main questions it aims to answer are:

if the anterior approach to the hip is faster recovery than lateral approach? if the anterior approach to the hip has better gait mechanics than lateral approach?

Participants will:

undergo one of the two approaches for total hip arthroplasty. All patients will be followed up at 2 weeks, 6 weeks, 3 months and 18 months. gait analysis will be done at 6wks, 3m, and 18months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary osteoarthritis or osteonecrosis of the hip who consented for treatment with a total hip arthroplasty (THA) through an anterior or lateral approach.
* Age between 20 - 60 years of age.
* The participant had to be independent and physically active, which characterized as having the capacity to carry out daily tasks, ascend two flights of stairs, and able to walk for 15 minutes.

Exclusion Criteria:

* Patients with bilateral hip affection.
* Body mass index (BMI) greater than 40.
* Diagnosis other than primary osteoarthritis or osteonecrosis.
* Prior hip or spine surgery.
* chronic uncontrolled comorbidities, psychological disorders.
* American Society of Anaesthesiologists score (ASA) higher than 2
* chronic neurological deficits that influence gait.
* any limb length discrepancy more than 1 cm.
* Any postoperative complication that will lead to delay in weight bearing.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
surgery time | intraoperative time starting from skin incision to skin closure
  by ''Minute'' as the unit, no special description.
hemoglobin drop | postoperative day one
  hemoglobin drop level between pre and postoperative.
hospital stays | immediately after the procedure
  by ''Day'' as the unit, no special description. postoperative stay days from operation day to discharge day.
pain score | 2 weeks 6 weeks 3 months 18 months
  using visual analogue scale (VAS) from 0-10 the more scale the worst the pain
Harris hip score | 2 weeks 6 weeks 3 months 18 months
  for measuring hip function from 0-100 the more the score the better hip function

SECONDARY OUTCOMES:
gait analysis | at 6 weeks, 3 months, 18 months
  A single experienced physical medicine specialist will perform the gait analysis in a gait lab. Three-dimensional kinematic and kinetic data will be collected using eight high-speed infrared cameras (Quality motion analysis system, oqus 1 cameras), which can capture 240 frames per second, two force plates (Advanced Mechanical Technology Incorporated, AMTI), and 26 ten-millimeter passive retroreflective markers fixed on the subject using a double-face tape in specific landmarks on the subject in accordance to the modified institute Orthopedic Rizzoli (IOR ) model for full body marker set.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasia, Egypt

REFERENCES:
- [Background] Wang Z, Bao HW, Hou JZ. Direct anterior versus lateral approaches for clinical outcomes after total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2019 Feb 26;14(1):63. doi: 10.1186/s13018-019-1095-z. PMID 30808382
- [Background] Pospischill M, Kranzl A, Attwenger B, Knahr K. Minimally invasive compared with traditional transgluteal approach for total hip arthroplasty: a comparative gait analysis. J Bone Joint Surg Am. 2010 Feb;92(2):328-37. doi: 10.2106/JBJS.H.01086. PMID 20124059
- [Background] Yue C, Kang P, Pei F. Comparison of Direct Anterior and Lateral Approaches in Total Hip Arthroplasty: A Systematic Review and Meta-Analysis (PRISMA). Medicine (Baltimore). 2015 Dec;94(50):e2126. doi: 10.1097/MD.0000000000002126. PMID 26683920
- [Background] Graves SC, Dropkin BM, Keeney BJ, Lurie JD, Tomek IM. Does Surgical Approach Affect Patient-reported Function After Primary THA? Clin Orthop Relat Res. 2016 Apr;474(4):971-81. doi: 10.1007/s11999-015-4639-5. Epub 2015 Nov 30. PMID 26620966
- [Background] Alecci V, Valente M, Crucil M, Minerva M, Pellegrino CM, Sabbadini DD. Comparison of primary total hip replacements performed with a direct anterior approach versus the standard lateral approach: perioperative findings. J Orthop Traumatol. 2011 Sep;12(3):123-9. doi: 10.1007/s10195-011-0144-0. Epub 2011 Jul 12. PMID 21748384
- [Background] Reichert JC, Volkmann MR, Koppmair M, Rackwitz L, Ludemann M, Rudert M, Noth U. Comparative retrospective study of the direct anterior and transgluteal approaches for primary total hip arthroplasty. Int Orthop. 2015 Dec;39(12):2309-13. doi: 10.1007/s00264-015-2732-8. Epub 2015 Mar 21. PMID 25795247
- [Background] Ilchmann T, Gersbach S, Zwicky L, Clauss M. Standard Transgluteal versus Minimal Invasive Anterior Approach in hip Arthroplasty: A Prospective, Consecutive Cohort Study. Orthop Rev (Pavia). 2013 Nov 6;5(4):e31. doi: 10.4081/or.2013.e31. eCollection 2013. PMID 24416475
- [Background] Yoo JI, Cha YH, Kim KJ, Kim HY, Choy WS, Hwang SC. Gait analysis after total hip arthroplasty using direct anterior approach versus anterolateral approach: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2019 Feb 8;20(1):63. doi: 10.1186/s12891-019-2450-2. PMID 30736783
- See also: Gait analysis after total hip arthroplasty using direct anterior approach versus anterolateral approach: a systematic review and meta-analysis — http://pubmed.ncbi.nlm.nih.gov/30736783/